CLINICAL TRIAL: NCT07223229
Title: A Phase 2, Randomized, Double-Blind, Placebo-controlled Proof-of-Concept Study to Evaluate the Efficacy and Safety of EI-001 in Patients With Nonsegmental Vitiligo
Brief Title: Phase 2 Study to Evaluate EI-001 in Non-segmental Vitiligo Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elixiron Immunotherapeutics (Hong Kong) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EI-001-201
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Non-segmental Vitiligo
MeSH Terms: interventions — BL-EI001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: EI-001 (Experimental)
  Interventions: Biological: EI-001
- Drug: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: EI-001 — EI-001 drug product is supplied as a colorless to slightly yellow and sterile solution for infusion with a protein concentration of 10.0 mg/mL
  Arms: Drug: EI-001
Other: Placebo — 0.9% sterile sodium chloride solution
  Arms: Drug: Placebo

SUMMARY:
The primary purpose of this study is to evaluate whether the drug EI-001 can help improve vitiligo symptoms. EI-001 is a novel antibody drug that affects the immune system to decrease uncontrolled inflammation. EI-001 has been investigated in human cell cultures, animal studies, and in a Phase 1 healthy volunteer study. The results so far show that EI-001 is a tolerable and potential new treatment for immune diseases such as vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the informed consent form (ICF).
* Male or female, aged 18-65 years at the time of consent.
* BMI 18-38 kg/m² and weight ≥ 40 kg at consent. Clinically diagnosed non-segmental vitiligo (NSV) for at least 3 months, and meets one of the following:
* Inadequate response to approved treatments:
* Topical therapy (e.g., corticosteroids, calcineurin inhibitors, or JAK inhibitors) ≥ 3 months,
* Phototherapy ≥ 6 months, or Oral therapy (e.g., corticosteroids, calcineurin inhibitors) ≥ 3 months.
* Or unable to use these treatments due to contraindications, intolerance, or unsuitability.
* Depigmentation extent meeting all of the following:

Facial BSA (F-BSA) ≥ 0.5%, Facial VASI (F-VASI) ≥ 0.5, Total BSA (T-BSA) between 5% and 60%, Total VASI (T-VASI) ≥ 5.

* Agree to discontinue all vitiligo treatments from screening until final follow-up.
* If not previously vaccinated against zoster, agree to complete vaccination before Day 1.
* Contraception
* Not applicable to females of non-childbearing potential (surgically sterile or postmenopausal ≥12 months, confirmed by FSH at screening).

Exclusion Criteria:

* Non-eligible skin conditions: Other types of vitiligo (e.g., segmental) or other depigmentation disorders (e.g., piebaldism, leprosy, post-inflammatory hypopigmentation, tinea versicolor, etc.), or ≥30% leukotrichia on face or body.
* Psychiatric risk
* Recent vitiligo treatments
* Surgical treatments or depigmenting agents (e.g., monobenzone)
* High-dose steroids
* Pregnancy or lactation
* Abnormal Medical conditions
* Prohibited prior therapies
* Cardiac abnormalities
* Abnormal chest X-ray
* Renal impairment
* Clinically significant abnormal laboratory results at screening, per investigator judgment.
* Viral infections:
* Hypersensitivity: Known allergy or severe reaction to EI-001 or its excipients.
* Compliance concerns: Any condition that would make it difficult for the subject to follow the study schedule, receive treatment, attend visits, or could interfere with study objectives, data interpretation, or participant safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in F-VASI from baseline | Week 24

SECONDARY OUTCOMES:
Proportion of subjects achieving F-VASI50 | Week 24
  F-VASI50 is defined as at least 50% improvement in F-VASI from baseline
Frequency and severity of AEs and SAEs | Week 32
  Including the results of physical examinations, vital signs, evaluation of clinical laboratory studies, and ECG
Absolute values and percent change in F-VASI from baseline at designated time points | Week 22
Absolute values and percent change in T-VASI from baseline at designated time points | Week 22
Proportion of subjects achieving F-VASI50/75, T-VASI50 at designated time points | Week 22
  F-VASI75 is defined as at least 75% improvement in F-VASI from baseline T-VASI50 is defined as at least 50% improvement in T-VASI from baseline

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Skin Care Research, LLC, Hollywood, Florida
  - U Mass Chan Medical School Department of Dermatology, Worcester, Massachusetts
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan